CLINICAL TRIAL: NCT02956642
Title: Study to Understand Gaining Access to Blood Glucose Records (SUGAR), A Randomized Controlled Trial of the Effect of the Livongo Health Diabetes Management Program vs. Standard Care on Glycemic Control
Brief Title: Study to Understand Gaining Access to Blood Glucose Records
Acronym: SUGAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Livongo Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EUR-001
Record Dates: First submitted 2016-10-31; First posted 2016-11-07 (Estimated); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Blood Glucose Monitoring System (Experimental): Participants in this arm will receive the Livongo Health System to manage diabetes. 150 participants will participate in this arm.
  Interventions: Device: Livongo Health System
- Standard Blood Glucose Monitoring (Active Comparator): Participants in this arm will receive the iHealth Glucose Meter to take blood glucose measurements that will then be compared to participants from the Livongo Health System arm. 150 participants will participate in this arm.
  Interventions: Device: iHealth Glucose Meter

INTERVENTIONS:
Device: Livongo Health System — Participants will be asked to use the Livongo Health System to manage their blood glucose.
  Arms: Blood Glucose Monitoring System
Device: iHealth Glucose Meter — Participants will be asked to use the iHealth Glucose Meter to take blood glucose measurements.
  Arms: Standard Blood Glucose Monitoring

SUMMARY:
This study is a two-arm randomized controlled trial in which participants will receive either the Livongo Health system or iHealth glucose meter for measuring their blood glucose. The study hypothesizes the use of the Livongo Health system results in a greater improvement in A1c compared to standard blood glucose monitoring, as demonstrated by the iHealth Bluetooth-enabled glucose meter.

DETAILED DESCRIPTION:
Participants in this study will partake in study surveys, daily blood glucose monitor measurements, and blood sampling for the duration of their participation. The study intends to recruit and randomize 300 participants.

1. Surveys and Measurements

   All study participants may complete surveys via their personal iOS smartphone device on: study qualification (intake survey/eligibility screener), diabetes status (initial diabetes survey), physical activity (iPAQ), quality of life (SF-12), vitals, demographics hospitalizations and interaction with health care provider (attached), and diabetes distress. Most survey data will be collected at 1, 3, and 6 months. There will also be Weekly Engagement surveys which will be two simple questions each week. At the end of the study, a Feedback survey will ask participants about their study experiences. Surveys will each have a simple description to introduce participants to the survey they are being asked to take. These surveys will be administered through the Eureka mHealth Research Platform, the study's main tool for data collection, data storage, and study management. Specific usability assessments that are native to the Livongo or iHealth platform may also be shown through the device to the participants in order to gather user feedback information.

   After qualifying and providing consent to participate in the study, participants will be referred to a convenient lab or receive a mail-in lab test kit for establishing hemoglobin A1c (A1c) levels and lipid panel levels. A1c tests will be collected at months 1 (baseline), 3, and 6 (closeout). For each A1c test performed in the lab, 1mL (milliliter) of blood will be drawn. Lipid panels (total cholesterol, LDL, HDL, and triglycerides) will be collected at months 1 (baseline) and 6 (closeout). For each lipid panel, 1mL of blood will be drawn. If participants elect to use a mail-in lab test kit, for each A1c test or lipid panel, 35 microliters of blood will be collected and mailed in for testing (total 75 microliters at months 1 and 6, and 30 microliters at month 3).
2. Randomization Once the baseline A1c value is obtained, the patient will be randomized (block randomization by diabetes type).
3. Device Usage After randomization, participants will receive either the Livongo Health system or the iHealth glucose meter by mail.

   If a participant is randomized to the iHealth treatment group, participants will download the iHealth iOS application and receive an iHealth blood glucose meter in the mail. Participants will link the iHealth application with a mobile version of the Eureka mHealth Research Platform.

   If a participant is randomized to the Livongo system treatment group, the participant will receive the Livongo blood glucose meter device in the mail, create a Livongo account, and link their Livongo account with the Eureka mHealth Research Platform. Livongo- or iHealth-specific instructions will be provided with each meter and a study coordinator will be available to answer study participant questions about using the BG meters. Participants may be referred to Livongo or iHealth customer service for technical support, if needed.

   Participants will not be given specific instructions on how often to check their BG, or how often they should use the Livongo system or iHealth glucose meter as a part of this study. This is done in order to determine the uptake of the intervention and resulting behavior without outside prompting.

   Participants will either use the Livongo system or the iHealth glucose meter for 6 months from the time of enrollment in the study.
4. Messaging/Reminders Participants who have been mailed a BG (Blood Glucose) meter but are not using the device after two weeks will be contacted by in-app push notifications, text messages, email or a phone call for device setup and/or assistance.

Participants will also receive reminders to complete study activities via in-app push notifications, text messages, email or a phone call.

Two weeks prior to the end of the study period, participants will be contacted by email and/or receive in-app push notifications to remind them to complete their A1c measurement and closeout surveys.

Note: Participation in this research study will not affect individual participants' standard clinical care for diabetes. Participants will remain under the care of their current health care provider and will be able to continue receiving all usual care from that provider. The health care provider will continue to provide recommendations for the number of times the participant should check their blood glucose. Although the participant wil be asked to use a different glucose meter for this study, the number of times they use it will still be determined by their health care provider. The same information that they received from their existing glucose meter will be available from the study glucose meter. During the study, they will be provided with glucose meter strips at no charge, to ensure that an insufficient number of strips will not interfere with their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* People with type 2 diabetes mellitus on any type of medication
* Adults, age 18 years or older
* iOS Smartphone with access to data and/or Wi-Fi
* Willing to answer survey questions throughout the study
* Willing to visit a lab for 3 blood draws at no cost to participants

Exclusion Criteria:

* Using continuous glucose monitoring during the study period
* Using an insulin pump during the study period
* Unable or unwilling to switch blood glucose meters to the study meter
* Hospitalization for Diabetic ketoacidosis (DKA) or hypoglycemia in the past 1 month prior to enrollment
* Pregnant patients, or intention to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenise Wong, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood Glucose Monitoring System | Standard Blood Glucose Monitoring
Started | 43 | 41
Completed | 42 | 38
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Glucose Monitoring System | Standard Blood Glucose Monitoring | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (11.6) | 60.5 (10.8) | 58.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 33 | 26 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 1 | 4
  Asian (including South Asian and Asian Indian) | 5 | 4 | 9
  Hispanic | 0 | 2 | 2
  non-Hispanic White | 35 | 34 | 69
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 41 | 84

OUTCOME MEASURES:

1. Primary Outcome: Mean HbA1c Levels
Description: Three HbA1c measures per study participant will be acquired at 3 points in the study duration (baseline, 3 months, and 6 months). In order to compare the changes in HbA1c, the values may be analyzed and separated with regard to duration of diabetes (days, months, years), and/or HbA1c levels at baseline. Reported in this table are the means for all participants for each given timepoint.
Time Frame: 6 months
Population: Of all study participants, 4 withdrew from the study (1 in the blood glucose monitoring system group, and 3 in the standard blood glucose monitoring group). The rest of the participants did not complete the lab draw activities and were lost to follow-up.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Groups:
- Blood Glucose Monitoring System: Participants in this arm will receive the Livongo Health System to manage diabetes.
  Livongo Health System: Participants will be asked to use the Livongo Health System to manage their blood glucose.
- Standard Blood Glucose Monitoring: Participants in this arm will receive the iHealth Glucose Meter to take blood glucose measurements that will then be compared to participants from the Livongo Health System arm.
  iHealth Glucose Meter: Participants will be asked to use the iHealth Glucose Meter to take blood glucose measurements.
Arm/Group | Blood Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 43 | 41
percentage of glycated hemoglobin
  Baseline | 8.0 (1.5) | 7.3 (1.1)
  3 months: number analyzed (Participants) | 31 | 29
  3 months | 7.9 (1.5) | 7.6 (1.2)
  6 months: number analyzed (Participants) | 20 | 24
  6 months | 7.9 (1.1) | 7.5 (1.1)

2. Primary Outcome: Change in HbA1c
Description: In this analysis, change in HbA1c within individual participants was compared from baseline to 6 months. Only participants with 6-month data were included.
Time Frame: 6 months
Population: This analysis included participants with data at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Blood Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 20 | 24
percentage of glycated hemoglobin | 0.31 (0.79) | 0.38 (0.83)

3. Secondary Outcome: Mean Fasting LDL
Description: As a secondary outcome, we will determine the effect of use of the Livongo Health system on fasting lipid panels (LDL). A lipid panel will be done at baseline, 3 months, and at 6 months. Reported in this table are means for all participants with data at each timepoint.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Blood Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 43 | 41
mg/dL
  Baseline | 81 (33.5) | 94.5 (26.7)
  3 months: number analyzed (Participants) | 31 | 29
  3 months | 73.9 (32) | 98.2 (51.7)
  6 months: number analyzed (Participants) | 20 | 24
  6 months | 87.9 (32.9) | 92.7 (48.8)

4. Secondary Outcome: Change in Fasting LDL
Description: In this analysis, change in fasting LDL within individual participants was compared from baseline to 6 months. Only participants with 6-month data were included.
Time Frame: 6 months
Population: This analysis included participants with data at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Blood Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 20 | 24
mg/dL | -0.3 (24.7) | -25.25 (35.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of participation in the study (6 months).
Arm/Group | Blood Glucose Monitoring System | Standard Blood Glucose Monitoring
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/41
Other Adverse Events (participants affected / at risk) | 0/43 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT02956642/Prot_SAP_000.pdf